CLINICAL TRIAL: NCT04165239
Title: A Phase IIb Double-blind, Randomised, Placebo-controlled, Multi-centre, Confirmative Three-way Cross-over Study on Cognitive Function With Two Doses of KH176 in Subjects With a Genetically Confirmed Mitochondrial DNA tRNALeu(UUR) m.3243A>G Mutation.
Brief Title: The KHENERGYZE Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khondrion BV (Industry)
Collaborators: Julius Clinical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH-176-202
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial Encephalomyopathies; MELAS Syndrome; MIDD
Keywords: Mitochondrial; Oxidative Phosphorylation (OXPHOS); MELAS; MIDD; KH176
MeSH Terms: conditions — Mitochondrial Diseases; Mitochondrial Myopathies; Mitochondrial Encephalomyopathies; MELAS Syndrome | interventions — 6-hydroxy-2,5,7,8-tetramethylchroman-2-carboxylic acid

STUDY DESIGN:
Intervention Model Description: The study will be a double-blind, randomised, placebo-controlled, multi-centre, three-way cross-over study. Twenty-seven subjects, with a confirmed mitochondrial DNA tRNALeu(UUR) 3243A>G mutation and with clinical signs of mitochondrial disease including attentional dysfunction, and fulfilling pre-defined cardiac exclusion criteria, will be randomised over three treatment sequences as assigned by Latin-square. Each group will have 3 treatment periods of 28 days each, separated by 14-day washout periods between treatments. During the 28-day treatment periods, subjects will receive bid oral administration of 50 mg KH176,100 mg KH176, or placebo in the sequence as applicable for the group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Oral administration of 50 mg KH176 twice daily
  Interventions: Drug: KH176
- Treatment B (Experimental): Oral administration of 100 mg KH176 twice daily
  Interventions: Drug: KH176
- Treatment C (Placebo Comparator): Oral administration of matching placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KH176 — Oral administration of 50 mg KH176 twice daily
  Other Names: Sonlicromanol
  Arms: Treatment A
Drug: KH176 — Oral administration of 100 mg KH176 twice daily
  Other Names: Sonlicromanol
  Arms: Treatment B
Drug: Placebo — Oral administration of matching placebo twice daily
  Arms: Treatment C

SUMMARY:
Mitochondrial diseases, estimated prevalence 1 in 4,300 adults, is caused by pathogenic mutations in genes finally encoding for mitochondrial proteins of the various enzyme complexes of the OXPHOS. Among these mutations, the 3243A>G nucleotide change in the mitochondrially encoded transfer RNALeu(UUR) leucine 1 gene (MT TL 1) is the most prevalent one. The OXPHOS dysfunction resulting from such mutations leads to increased production of reactive oxygen species (ROS), ultimately leading to irreversible oxidative damage of macromolecules, or to more selective and reversible redox modulation of cell signaling that may impact (adult) neurogenesis.

Despite advances in the understanding of mitochondrial disorders, treatment options are extremely limited and, to date, largely supportive. Therefore, there is an urgent need for novel treatments. KH176, a new active pharmaceutical ingredient (API), is an orally bio-available small molecule under development for the treatment of these disorders (see Section 1.4). The current study will further evaluate the effect of KH176 in various cognitive domains and evaluate the effect of different doses of KH176 (See Section 1.5).

In view of the growing recognition of the importance of mitochondrial function in maintaining cognitive processes in the brain, as well as the understanding of the safety profile and pharmacokinetics of KH176 following the two clinical studies described above, a more detailed study is indicated of the effects of KH176 in various cognitive domains, using the confirmed safe and well-tolerated KH176 dose of 100 mg bid, as well as a lower dose of 50 mg bid. The primary objective is an evaluation of KH176 in the attention domain of cognitive functioning, as assessed by the visual identification test score of the Cogstate computerised cognitive testing battery.

DETAILED DESCRIPTION:
For this study, a 3 x 3 crossover design will be applied, i.e., with 3 treatments, 3 sequences and 3 periods, employing a Latin square assignment. Using this design, each subject will function as his/her own control. This will reduce variability and thus increase the chances of observing true effects between treatment periods (effects of treatment compared to placebo). In each treatment period, assessments will be performed at baseline prior to dosing and post dosing, enabling a change from baseline analysis and enabling the possibility to compare baseline conditions for each treatment period. The treatment period in each treatment is 28 days (4 weeks), which is supported by the pre-clinical toxicology program. In mouse studies, a 4-week period was sufficient to observe clinically relevant effects.

ELIGIBILITY:
1. Males and females aged 18 years or older at screening.
2. Ability and willingness to provide written Informed Consent prior to screening evaluations.
3. Confirmed mitochondrial DNA tRNALeu(UUR) m.3243A>G mutation.
4. Positive NMDAS score >10 at Screening.
5. Three or more clinical features, with no other causative unifying diagnosis, found to commonly occur in subjects with a m.3243A>G mutation:

   * Deafness
   * Developmental delay
   * Diabetes Mellitus
   * Epilepsy
   * Gastrointestinal complaints
   * Progressive External Ophtalmoplegia (PEO) and retinopathy
   * Ataxia
   * Exercise intolerance
   * Fatigue
   * Migraine (with or without aura), specified by at least five attacks fulfilling diagnostic criteria B-D:

B. Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)

C. Headache has at least two of the following four characteristics:

1. unilateral location
2. pulsating quality
3. moderate or severe pain intensity
4. aggravation or causing avoidance of routine physical activity (e.g. walking or climbing stairs)

D. During headache at least one of the following:

1. nausea and/or vomiting 2. photophobia and phonophobia 6. Attentional dysfunction score (Cogstate Identification test) ≥ 0.5 standard deviations poorer than healthy controls at Screening.

7. Disease appropriate physical and mental health as established at Screening by medical history, physical examination, ECG and vital signs recording, and results of clinical chemistry and haematology testing as judged by the investigator.

8. Objectified Left Ventricular Ejection Fraction (LVEF) ≥45% (echocardiography, or otherwise).

9. Left Ventricular (LV) wall thickness ≤15 mm. 10. Left atrium dilatation ≤ 40 mL/m2. Note: No need to test LV parameters (criteria #8, #9, #10) if favourable echocardiography (or otherwise) results dated less than 6 months prior to Screening are available.

11. Women of childbearing potential must be willing to use highly effective contraceptive methods during the entire study, i.e., combined (estrogen and progestogen containing) oral, intravaginal or transdermal hormonal contraception associated with inhibition of ovulation;, oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation; use of an intrauterine device; an intrauterine hormone releasing system, bilateral tubal occlusion and vasectomy of the partner.

Any hormonal contraception method must be supplemented with a barrier method (preferably male condom).

Vasectomised partner is considered a highly effective birth control method provided that partner is the sole sexual partner of the subject and that the vasectomised partner has received medical assessment of the surgical success. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. Reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Note 1: Natural family planning methods, female condom, cervical cap or diaphragm are not considered adequate contraceptive methods in the context of this study.

Note 2: To be considered not of childbearing potential, potential female subjects must be post-menopausal for at least two years, or have been surgically sterilised (bilateral tubal ligation, hysterectomy or bilateral oophorectomy) for at least 6 months prior to Screening.

Note 3: KH176 has been shown non-genotoxic judged from the Ames test, Chromosomal Aberration test and in vivo Micronucleus test. Moreover, appreciable systemic exposure from the exposure to (~2.5 mL) semen is extremely unlikely. However, until reproductive toxicology studies have confirmed that KH176 does not adversely affect normal reproduction in adult males and females, as well as causing developmental toxicity in the offspring, the following contraceptive precautions must be adhered to:

* male subjects with female partners of childbearing potential must be willing to use condoms during the entire study.
* female partners of childbearing potential of male subjects must be willing to use adequate contraceptive methods during the entire study, i.e., a hormonal contraceptive method (pill, vaginal ring, patch, implant, injectable, hormone-medicated intrauterine device) or an intrauterine device.

  12. Able to comply with the study requirements, including swallowing study medication.

Exclusion Criteria

1. Surgery of gastro-intestinal tract that might interfere with absorption.
2. Treatment with an investigational product within 3 months or 5 times the half-life of the investigational product (whichever is longer) prior to the first dose of the study medication.
3. Documented history of ventricular tachycardia (HR>110 beats/min).
4. History of acute heart failure, (family) history of unexplained syncope or congenital long and short QT syndrome or sudden death.
5. Clinically relevant abnormal laboratory, vital signs or physical or mental health;

   1. Aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) > 3 x upper limit of normal (ULN), or bilirubin > 3 x ULN at screening. If a patient has ASAT or ALAT > 3 x ULN but < 3.5 x ULN, re-assessment is allowed at the investigator's discretion.
   2. Estimated glomerular filtration rate ≤ 60 mL/min according to the CKD-EPI formula at screening.
   3. Systolic Blood pressure > 150 mmHg at screening or baseline.
   4. All other clinically relevant parameters at screening or baseline as judged by the Investigator.
6. Clinically relevant abnormal ECG or cardiac functioning, defined as ST-segment elevation > 1 mm in I, II, III, aVL ,aVF ,V3 ,V4 ,V5 ,V6; > 2 mm in V1, V2; QTc > 450 ms for male subjects; QTc: > 470ms for female subjects (local, machine read), T-top inversion in >1 consecutive lead.
7. Serum Hyper-potassium (> 5.0 mEq/L).
8. Serum Hypo-potassium (< 3.5 mEq/L).
9. History of ischemic heart disease.
10. Symptomatic heart failure.
11. Clinically relevant aorta and/or mitralis valvular defect as judged by the investigator.
12. Pregnancy or breast feeding (females).
13. Poor nutritional state as judged by the investigator.
14. History of hypersensitivity or idiosyncrasy to any of the components of the investigational drug.
15. Medical history of drug abuse (illegal drugs such as cannabinoids, amphetamines, cocaine, opiates or problematic use of prescription drugs such as benzodiazepines, opiates).
16. The use of any of the following medication and/or supplements within 4 weeks or 5 times the half-life (whichever is longer) prior to the first dosing of the study medication:

    1. (multi)vitamins, co-enzyme Q10, Vitamin E, riboflavin, and anti-oxidant supplements (including, but not limited to idebenone/EPI-743, mitoQ); unless stable for at least one month before first dosing and remaining stable throughout the study.
    2. any medication negatively influencing mitochondrial functioning (including but not limited to valproic acid, glitazones, statins, anti-virals, amiodarone, and non-steroidal anti-inflammatory drugs (NSAIDs)), unless stable for at least one month before first dosing and remaining stable throughout the study.

       Note: thus, mitoQ and any medication negatively influencing mitochondrial functioning are allowed as long as the dose has been stable for at least one month prior to first dosing and remains stable throughout the study.
    3. any strong Cytochrome P450 (CYP)3A4 inhibitors (all 'conazoles-anti-fungals', HIV antivirals, grapefruit).
    4. strong CYP3A4 inducers (including HIV antivirals, carbamazepine, phenobarbital, phenytoin, rifampicin, St. John's wort, pioglitazone, troglitazone).
    5. any medication known to affect cardiac repolarisation, unless the QTc interval at screening is normal during stable treatment (all anti-psychotics, several anti-depressants, e.g. nor/amitriptyline, fluoxetine, anti-emetics: domperidone (motilium®) granisetron, ondansetron). For a complete list see https://crediblemeds.org.
    6. any medication metabolised by CYP with a narrow therapeutical width. For reference (Germany and United Kingdom): drug interaction table of Indiana University (http://medicine.iupui.edu/clinpharm/ddis/clinical-table/). For reference (The Netherlands): KNMP Kennisbank (https://www.knmp.nl/producten/knmp-kennisbank/inloggen-knmp-kennisbank. For reference (all other countries): drug interaction table of Indiana University (http://medicine.iupui.edu/clinpharm/ddis/clinical-table/).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning: Attention | One month
  The attention domain score of cognitive functioning, as assessed by the visual Identification Test of the Cogstate computerised cognitive testing battery

SECONDARY OUTCOMES:
Executive functioning | One month
  The executive functioning domain score of cognitive functioning, as assessed by the Groton Maze Learning Test of the Cogstate computerised cognitive testing battery
Psychomotor function | One month
  The psychomotor functioning domain score of cognitive functioning, as assessed by the Detection Test of the Cogstate computerised cognitive testing battery
Working Memeory | One month
  The working memory domain score of cognitive functioning, as assessed by the One Back Test of the Cogstate computerised cognitive testing battery
Visual learning | One month
  The visual learning domain score of cognitive functioning, as assessed by the One Card Learning Test of the Cogstate computerised cognitive testing battery
Verbal learning | One month
  The verbal learning functioning domain score of cognitive functioning, as assessed by the International Shopping List Test of the Cogstate computerised cognitive testing battery
Test of Attentional Performance (TAP) | One month
  Standardised test to evaluate alertness and mental flexibility
Beck Depression Inventory | One month
  21-question multiple-choice self-report inventory, for measuring the severity of depression
Hamilton Anxiety and Depression Score (HADS) | One month
  Subject-reported outcome measure and comprises 14 items equally divided over the two subscales anxiety (HADS-A) and depression (HADS-D)
Newcastle Mitochondrial Disease Scale for Adults (NMDAS) | One month
  Semi-quantitative clinical rating scale designed for mitochondrial disease. The rating scale explores several domains: current function, system specific involvement, current clinical assessment and quality of life
Number of headache days | One month
  Self report diary
Pure Tone Audiometry (PTA) | One month
  Standardized test measure individual hearing threshold levels
University of Penn Smell Identification Test (UPSIT) | One month
  Test to measure the individual's ability to detect odors at a suprathreshold level.
Cognitive Failure Questionnaire (CFQ) | One month
  Questionnaire to evaluate subjective cognitive functioning.
Neuro-QoL Fatigue Short Form (quality in life in neurological disorders) | One month
  8-item self assessment questionnaire evaluating the perception of fatigue and its impact in daily life activities

CONTACTS AND LOCATIONS:
Locations (4):
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- Friedrich-Baur Institut, München, Bavaria, Germany
- Radboud University Medical Center, Nijmegen, Netherlands
- Institute for Ageing and Health Newcastle University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No